CLINICAL TRIAL: NCT02979444
Title: Comparing the Effectiveness of Clinicians and Paraprofessionals to Reduce Disparities in Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Darius Tandon, Associate Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STU00203761
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Perinatal Depression; PostPartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mothers and Babies Groups Home-Visitor (Experimental): Women who participate in the home-visitor led arm will receive the intervention from a paraprofessional home-visitor and complete assessments at baseline, post-intervention, and 12 and 24 weeks postpartum.
  Interventions: Behavioral: Mothers and Babies Groups
- Mothers and Babies Groups Clinician (Experimental): Women who participate in the mental health consultant led arm will receive the intervention from a mental health consultant and complete assessments at baseline, post-intervention, and 12 and 24 weeks postpartum.
  Interventions: Behavioral: Mothers and Babies Groups
- Control (No Intervention): Women who participate in the control arm will not receive the intervention but will complete assessments at baseline, 8 weeks post-baseline, and 12 and 24 weeks postpartum.

INTERVENTIONS:
Behavioral: Mothers and Babies Groups — The Mothers and Babies group intervention is comprised of 6, two hour sessions. It is divided into three overall sections, one on each of the following Cognitive Behavioral Theory components; Pleasant Activities, Thoughts, and Contact with Others. In each of these sections, participants are first taught to understand how the component influences her mood. This teaching of the relationships between CBT components and mood is referred to as psychoeducation. In addition to psychoeducation, participants also receive concrete skills in each of the three sections (pleasant activities, thoughts, contact with others). These skills are intended to provide participants with a "toolkit" of approaches they can use to improve their mood.
  Arms: Mothers and Babies Groups Clinician; Mothers and Babies Groups Home-Visitor

SUMMARY:
There is considerable evidence that most perinatal women at risk for postpartum depression do not engage in mental health services, even when referred by home visiting (HV) programs, primary care physicians, obstetricians, or gynecologists. Thus, interventions that can be delivered via alternative settings-e.g., HV programs-are essential to prevent the onset of major depression and worsening of depressive symptoms among perinatal women. This Patient Centered Outcomes Research Institute (PCORI) funded project aims to evaluate whether the Mothers and Babies (MB) group intervention, when led by paraprofessional home visitors, is more efficacious than usual care (i.e., home visiting without the MB enhancement). It will also examine if MB, when led by paraprofessional home visitors, is not inferior to MB delivered by mental health professionals. The results of this study will inform decision-making by HV programs regarding provision of MB to perinatal women at risk for developing major depression.

DETAILED DESCRIPTION:
Study Aims:

Aim #1 is to conduct a superiority trial that compares the efficacy of MB delivered by paraprofessional home visitors versus usual care (i.e., home visiting without MB) on patient-reported outcomes, including depressive symptoms, quality of life, parenting practices, engagement in pleasant activities, and relationship with one's partner.

Aim #2 is to conduct a non-inferiority trial that compares the effectiveness of MB delivered by (a) mental health clinicians versus (b) paraprofessional home visitors.

Aim #3 is to evaluate whether effectiveness of the two versions of MB (clinician led vs. paraprofessional home visitor led) varies according to patient characteristics (e.g., race, ethnicity, first-time mother, and/or geographic type of home visiting (HV) program (i.e., urban vs. rural).

Aim #4 is to examine the feasibility and acceptability of MB delivered by paraprofessional home visitors and mental health clinicians.

Postpartum depression is a serious mental health disorder that poses significant health and mental health risks for mothers and their infants. Research suggests that prevalence rates of postpartum depression are higher among low-income women than among middle-or high-income women. There is also consistent evidence that low-income women are less likely to receive mental health services in the perinatal (i.e., pregnancy until child's first birthday) period than their more affluent counterparts due to a variety of factors including stigma related to mental health service use and lack of access to community-based mental health providers. Postpartum depression is a particularly serious problem for low-income women, as it has the potential to create two generations of suffering, for both mother and child. It is estimated that over 10% of low-income infants have a mother who has major depression and more than 50% have a mother with some depressive symptoms. Postpartum depression has negative consequences for maternal parenting practices. Compared with women not suffering from postpartum depression, depressed women tend to be less positive, less spontaneous, and less responsive with their infants. Postpartum depression has been linked to developmental delays among infants of depressed mothers, including social interaction difficulties, attachment insecurity, and cognitive impairments.

Home visiting (HV) programs that provide services to perinatal women are one of the largest avenues through which perinatal women come to the attention of service providers, making HV a unique and viable setting for delivering mental health services. Although professional HV models exist (e.g., Nurse-Family Partnership), most HV programs in the United States use paraprofessionals. Previously, study investigators have established the efficacy of a group-based intervention -the Mothers and Babies (MB) Course-in preventing the onset of postpartum depression and reducing depressive symptoms when led by mental health professionals. However, to date there are no interventions led by non-health or non-mental health professionals that have demonstrated efficacy in preventing the onset and worsening of postpartum depression among low-income women. This project attempts to fill this notable gap.

The investigators will conduct a cluster randomized trial in which HV clients receive either a) MB delivered by mental health professionals, b) MB delivered by paraprofessional home visitors, or c) usual home visiting services. This study design will allow the investigators to conduct a superiority trial that compares the efficacy of MB delivered by paraprofessional home visitors versus usual care. A superiority trial will allow the investigators to generate efficacy data on MB delivered by paraprofessional home visitors. The study design will also allow the investigators to conduct a non-inferiority trial that compares the effectiveness of MB delivered by mental health professionals versus paraprofessional home visitors. Should the investigators find that paraprofessional home visitors are not inferior to mental health professionals in delivering the intervention, HV programs throughout the United States will be able to implement the MB Course with paraprofessional home visitors-an approach that is considerably more efficient and cost-effective than employing mental health professionals.

This study was born out of community stakeholders' need and desire for a low-cost intervention that could prevent the onset and worsening of depression among low-income women enrolled in HV programs. Maternal depression is an enormous challenge facing HV programs. However, there is consistent evidence that low-income women exhibiting depressive symptoms-including women enrolled in HV programs-do not access mental health treatment in the community. Lack of available mental health professionals, stigma in seeking mental health services, and logistical challenges (e.g., childcare, transportation) are a few of the barriers faced by perinatal women seeking mental health services. For those clients who do access services, most perinatal women are likely to receive pharmacological treatments, despite the fact that the vast majority of perinatal women prefer non-pharmacologic interventions.

HV programs are ideal settings for delivering mental health care to perinatal women because their mission is not stigmatizing and HV programs tend to be trusted entities in the communities they serve. However, there is not yet an evidence-based intervention that can be delivered by paraprofessionals (such as home visitors), thereby limiting HV programs' capacity to meet the needs of their clients needing mental health services.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will enroll only pregnant women in this study, given that the Mothers and Babies Course is delivered prenatally as a postpartum depression prevention intervention. The investigators will offer participation to prenatal home visiting clients, ages 16 and older, knowing the client base for home visiting programs includes pregnant teens.

Exclusion Criteria:

* Women with high-risk medical and pregnancy conditions will be excluded since this may preclude women from regularly attending intervention sessions. The investigators will not exclude women based on race/ethnicity or based on demographic characteristics other than the ability to speak English or Spanish.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 874 (Actual)
Dates: Start 2016-08; Primary Completion 2019-08-05 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darius Tandon, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams LS, Dornig K, Curran L. Barriers to service use for postpartum depression symptoms among low-income ethnic minority mothers in the United States. Qual Health Res. 2009 Apr;19(4):535-51. doi: 10.1177/1049732309332794. PMID 19299758
- [Background] Catanzaro SJ, Mearns J. Measuring generalized expectancies for negative mood regulation: initial scale development and implications. J Pers Assess. 1990 Summer;54(3-4):546-63. doi: 10.1080/00223891.1990.9674019. PMID 2348341
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Fresco DM, Moore MT, van Dulmen MH, Segal ZV, Ma SH, Teasdale JD, Williams JM. Initial psychometric properties of the experiences questionnaire: validation of a self-report measure of decentering. Behav Ther. 2007 Sep;38(3):234-46. doi: 10.1016/j.beth.2006.08.003. Epub 2007 Apr 24. PMID 17697849
- [Background] Gaynes BN, Gavin N, Meltzer-Brody S, Lohr KN, Swinson T, Gartlehner G, Brody S, Miller WC. Perinatal depression: prevalence, screening accuracy, and screening outcomes. Evid Rep Technol Assess (Summ). 2005 Feb;(119):1-8. doi: 10.1037/e439372005-001. No abstract available. PMID 15760246
- [Background] Grace SL, Evindar A, Stewart DE. The effect of postpartum depression on child cognitive development and behavior: a review and critical analysis of the literature. Arch Womens Ment Health. 2003 Nov;6(4):263-74. doi: 10.1007/s00737-003-0024-6. PMID 14628179
- [Background] Huybrechts KF, Palmsten K, Mogun H, Kowal M, Avorn J, Setoguchi-Iwata S, Hernandez-Diaz S. National trends in antidepressant medication treatment among publicly insured pregnant women. Gen Hosp Psychiatry. 2013 May-Jun;35(3):265-71. doi: 10.1016/j.genhosppsych.2012.12.010. Epub 2013 Jan 30. PMID 23374897
- [Background] Leis JA, Mendelson T, Perry DF, Tandon SD. Perceptions of mental health services among low-income, perinatal African-American women. Womens Health Issues. 2011 Jul-Aug;21(4):314-9. doi: 10.1016/j.whi.2011.03.005. PMID 21712144
- [Background] Meijer JL, Beijers C, van Pampus MG, Verbeek T, Stolk RP, Milgrom J, Bockting CL, Burger H. Predictive accuracy of Edinburgh postnatal depression scale assessment during pregnancy for the risk of developing postpartum depressive symptoms: a prospective cohort study. BJOG. 2014 Dec;121(13):1604-10. doi: 10.1111/1471-0528.12759. Epub 2014 Apr 7. PMID 24703235
- [Background] Rich-Edwards JW, Kleinman K, Abrams A, Harlow BL, McLaughlin TJ, Joffe H, Gillman MW. Sociodemographic predictors of antenatal and postpartum depressive symptoms among women in a medical group practice. J Epidemiol Community Health. 2006 Mar;60(3):221-7. doi: 10.1136/jech.2005.039370. PMID 16476752
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Sohr-Preston SL, Scaramella LV. Implications of timing of maternal depressive symptoms for early cognitive and language development. Clin Child Fam Psychol Rev. 2006 Mar;9(1):65-83. doi: 10.1007/s10567-006-0004-2. PMID 16817009
- [Background] Trivedi MH, Rush AJ, Ibrahim HM, Carmody TJ, Biggs MM, Suppes T, Crismon ML, Shores-Wilson K, Toprac MG, Dennehy EB, Witte B, Kashner TM. The Inventory of Depressive Symptomatology, Clinician Rating (IDS-C) and Self-Report (IDS-SR), and the Quick Inventory of Depressive Symptomatology, Clinician Rating (QIDS-C) and Self-Report (QIDS-SR) in public sector patients with mood disorders: a psychometric evaluation. Psychol Med. 2004 Jan;34(1):73-82. doi: 10.1017/s0033291703001107. PMID 14971628
- [Background] van Doesum KTM, Hosman CMH, Riksen-Walraven JM, Hoefnagels C. Correlates of depressed mothers' sensitivity toward their infants: the role of maternal, child, and contextual characteristics. J Am Acad Child Adolesc Psychiatry. 2007 Jun;46(6):747-756. doi: 10.1097/CHI.0b013e318040b272. PMID 17513987
- [Background] Zittel-Palamara K, Rockmaker JR, Schwabel KM, Weinstein WL, Thompson SJ. Desired assistance versus care received for postpartum depression: access to care differences by race. Arch Womens Ment Health. 2008 Jun;11(2):81-92. doi: 10.1007/s00737-008-0001-1. Epub 2008 May 8. PMID 18463943
- [Background] Kanter, J.W., Mulick, P.S., Busch, A.M., Berlin, K.S., & Martell, C.R. (2007). The Behavioral Activation for Depression Scale (BADS): Psychometric properties and factor structure. Journal of Psychopathology and Behavioral Assessment, 29, 191-202.
- [Background] Kanter, J.W., Rusch, L.C., Busch, A.M., & Sedivy, S.K. (2009). Validation of the behavioral activation for depression scale (BADS) in a community sample with elevated depressive symptoms. Journal of Psychopathology and Behavioral Assessment, 31, 36-42.
- [Background] Teri L, Lewinsohn P. Modification of the Pleasant and Unpleasant Events Schedules for use with the elderly. J Consult Clin Psychol. 1982 Jun;50(3):444-5. doi: 10.1037//0022-006x.50.3.444. No abstract available. PMID 7096747
- [Background] O'Hara, M., & Swain, A. (1996). Rates and risk of postpartum depression: A meta-analysis. International Review of Psychiatry, 8, 37-54.
- [Derived] Tandon SD, Johnson JK, Diebold A, Segovia M, Gollan JK, Degillio A, Zakieh D, Yeh C, Solano-Martinez J, Ciolino JD. Comparing the effectiveness of home visiting paraprofessionals and mental health professionals delivering a postpartum depression preventive intervention: a cluster-randomized non-inferiority clinical trial. Arch Womens Ment Health. 2021 Aug;24(4):629-640. doi: 10.1007/s00737-021-01112-9. Epub 2021 Mar 3. PMID 33655429
- [Derived] Diebold A, Segovia M, Johnson JK, Degillio A, Zakieh D, Park HJ, Lim K, Tandon SD. Acceptability and appropriateness of a perinatal depression preventive group intervention: a qualitative analysis. BMC Health Serv Res. 2020 Mar 7;20(1):189. doi: 10.1186/s12913-020-5031-z. PMID 32143644
- [Derived] Ciolino JD, Diebold A, Jensen JK, Rouleau GW, Koloms KK, Tandon D. Choosing an imbalance metric for covariate-constrained randomization in multiple-arm cluster-randomized trials. Trials. 2019 May 28;20(1):293. doi: 10.1186/s13063-019-3324-5. PMID 31138319
- [Derived] Jensen JK, Ciolino JD, Diebold A, Segovia M, Degillio A, Solano-Martinez J, Tandon SD. Comparing the Effectiveness of Clinicians and Paraprofessionals to Reduce Disparities in Perinatal Depression via the Mothers and Babies Course: Protocol for a Cluster-Randomized Controlled Trial. JMIR Res Protoc. 2018 Nov 20;7(11):e11624. doi: 10.2196/11624. PMID 30459138

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were randomized to one of the three study arms
Groups:
- Mothers and Babies Groups Home-Visitor: Women who participate in the home-visitor led arm will receive the intervention from a paraprofessional home visitor and complete assessments at baseline, post-intervention, and 12 and 24 weeks postpartum.
  Mothers and Babies Groups: The Mothers and Babies group intervention is comprised of 6, two hour sessions. It is divided into three overall sections, one on each of the following Cognitive Behavioral Theory components: Pleasant Activities, Thoughts, and Contact with Others. In each of these sections, participants are first taught to understand how the component influences her mood. This teaching of the relationships between CBT components and mood is referred to as psychoeducation. In addition to psychoeducation, participants also receive concrete skills in each of the three sections (pleasant activities, thoughts, contact with others). These skills are intended to provide participants with a "toolkit" of approaches they can use to improve their mood.
- Mothers and Babies Groups Clinician: Women who participate in the mental health consultant led arm will receive the intervention from a mental health consultant and complete assessments at baseline, post-intervention, and 12 and 24 weeks postpartum.
  Mothers and Babies Groups: The Mothers and Babies group intervention is comprised of 6, two hour sessions. It is divided into three overall sections, one on each of the following Cognitive Behavioral Theory components: Pleasant Activities, Thoughts, and Contact with Others. In each of these sections, participants are first taught to understand how the component influences her mood. This teaching of the relationships between CBT components and mood is referred to as psychoeducation. In addition to psychoeducation, participants also receive concrete skills in each of the three sections (pleasant activities, thoughts, contact with others). These skills are intended to provide participants with a "toolkit" of approaches they can use to improve their mood.
- Control: Women who participate in the control arm will not receive the intervention but will complete assessments at baseline, 8 weeks post-baseline, and 12 and 24 weeks postpartum. These women will receive usual home visiting services.
Period: Overall Study
Arm/Group | Mothers and Babies Groups Home-Visitor | Mothers and Babies Groups Clinician | Control
Started | 405 | 310 | 159
Completed | 382 | 293 | 149
Not Completed | 23 | 17 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mothers and Babies Groups Home-Visitor | Mothers and Babies Groups Clinician | Control | Total
Number analyzed (Participants) | 405 | 310 | 159 | 874
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.42 (5.82) | 25.80 (6.01) | 25.81 (5.39) | 26.09 (5.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405 | 310 | 159 | 874
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black/African American | 229 | 129 | 24 | 382
  Race/Ethnicity: White | 76 | 82 | 99 | 257
  Race/Ethnicity: Hispanic/Latina | 63 | 79 | 24 | 166
  Race/Ethnicity: Asian American | 2 | 3 | 4 | 9
  Race/Ethnicity: Native American | 5 | 1 | 0 | 6
  Race/Ethnicity: Biracial | 19 | 8 | 6 | 33
  Race/Ethnicity: Unknown | 11 | 8 | 2 | 21
Region of Enrollment [Number; unit: participants]
  United States | 405 | 310 | 159 | 874

OUTCOME MEASURES:

1. Primary Outcome: The Change in QIDS-16 Scores From Baseline to 24 Weeks Postpartum
Description: Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR16). The QIDS-SR16 was used to assess severity of depressive symptoms consistent with Diagnostic and Statistical Manual symptom criteria. Total scores range from 0-27; higher scores indicate greater symptomatology. The investigators anticipate a clinically meaningfully difference to be on the order of five points (as this is the difference in score on each severity level of depression) (Trivedi et al., 2004). For our non-inferiority analyses comparing MB led by home visitors vs. MB led by mental health clinicians, we will have >85% power to detect a difference difference in mean QIDS-16 scores of two points between the two active intervention arms.
Time Frame: Baseline and 12 and 24-week postpartum follow-up
Population: These numbers reflect the number of study participants with complete data at our 24-week postpartum assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mothers and Babies Groups Home-Visitor | Mothers and Babies Groups Clinician | Control
Number analyzed (Participants) | 365 | 272 | 146
score on a scale
  24-Week Postpartum Time Point | 5.9 (4.5) | 5.3 (4.5) | 5.8 (4.6)
  12- Week Postpartum Time Point | 6.4 (4.5) | 5.5 (4.5) | 5.9 (4.1)
  Baseline | 8.6 (4.3) | 7.8 (4.3) | 6.7 (3.6)

2. Secondary Outcome: The Change in the Behavioral Activation Scale From Baseline to 24-weeks Postpartum
Description: Behavioral Activation will be measured using the Behavioral Activation Depression Scale (BADS). The BADS assesses behaviors hypothesized to underlie depression and specifically targeted for change by behavioral activation strategies. It examines changes in the following areas: activation, avoidance/ rumination, work/school impairment, and social impairment. The BADS consists of 25 items, each rated on a seven point scale ranging from 0 (not at all) to 6 (completely). The range of the scale is 0-64. For the total scale, higher scores represent increased activation. The BADS has demonstrated strong internal consistency, construct validity, and predictive validity (Kanter et al, 2007; Kanter et al., 2009).
Time Frame: Baseline and 12 and 24-week postpartum follow-ups
Population: Overall number of participants analyzed at 24-weeks postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mothers and Babies Groups Home-Visitor | Mothers and Babies Groups Clinician | Control
Number analyzed (Participants) | 365 | 272 | 146
score on a scale
  24-Week Postpartum Time Point | 3.6 (1.1) | 3.8 (1.1) | 4.0 (1.1)
  12- Week Postpartum Time Point | 3.6 (1.1) | 3.8 (1.1) | 4.1 (1.1)
  Baseline | 3.6 (1.1) | 3.8 (1.1) | 4.1 (1.1)

3. Secondary Outcome: The Change in the Negative Mood Regulation Scale
Description: Mood regulation will be measured using the 30-item Negative Mood Regulation Scale (NMRS) (Catanzaro & Means, 1990). For each question, respondents use a 5-point scale to indicate what they believe they can do when they are disappointed or experiencing a negative mood. For our analyses, these items were averaged to create a mean NMRS score (range 1-5). Higher scores indicate a greater ability to regulate one's mood.
Time Frame: Baseline and 12 and 24-week postpartum follow-ups
Population: Participants analyzed at 24-weeks postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mothers and Babies Groups Home-Visitor | Mothers and Babies Groups Clinician | Control
Number analyzed (Participants) | 365 | 272 | 146
score on a scale
  24-Week Postpartum Time Point | 3.7 (0.6) | 3.8 (0.6) | 3.8 (0.7)
  12- Week Postpartum Time Point | 3.7 (0.6) | 3.8 (0.6) | 3.9 (0.6)
  Baseline | 3.6 (0.6) | 3.7 (0.6) | 3.9 (0.6)

4. Secondary Outcome: The Change in the MOS Social Support Survey From Baseline to 24-Weeks Postpartum
Description: Social support will be measured using the 19-item Medical Outcomes Study Social Support Survey (MOS-SSS) (Sherbourne & Stewart, 1991). This brief self-administered survey includes an overall functional social support index, as well as four functional support subscales: affectionate, emotional/informational, tangible, and positive social interaction. The range is 1-5 with greater scores indicating more perceived social support.
Time Frame: Baseline and 12 and 24-week follow-ups
Population: Participants analyzed at the 24-week postpartum time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mothers and Babies Groups Home-Visitor | Mothers and Babies Groups Clinician | Control
Number analyzed (Participants) | 365 | 272 | 146
score on a scale
  24-Week Postpartum Time Point | 3.8 (1.2) | 3.8 (1.1) | 4.1 (1.0)
  12- Week Postpartum Time Point | 3.8 (1.1) | 3.9 (1.2) | 4.2 (1.0)
  Baseline | 3.6 (1.2) | 3.7 (1.2) | 4.2 (1.0)

5. Secondary Outcome: The Change in the Experiences Questionnaire From Baseline to 24-Weeks Postpartum
Description: Decentering will be measured using the Experiences Questionnaire (EQ) (Fresco et al., 2007). The EQ is a 20 item self-report scale designed to measure decentering and rumination, which has demonstrated strong internal consistency in a number of studies examining effects of interventions that incorporate cognitive restructuring techniques. Response choices are on a 1-5 scale. For the purposes of our analyses, we created a mean EQ score (range 1-5), with higher scores indicating more decentering/rumination.
Time Frame: Baseline and 12 and 24-week follow-ups
Population: Participants analyzed at 24-weeks postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mothers and Babies Groups Home-Visitor | Mothers and Babies Groups Clinician | Control
Number analyzed (Participants) | 365 | 272 | 146
score on a scale
  24-Week Postpartum Time Point | 3.4 (0.8) | 3.5 (0.7) | 3.5 (0.7)
  12- Week Postpartum Time Point | 3.4 (0.7) | 3.4 (0.8) | 3.5 (0.6)
  Baseline | 3.4 (0.7) | 3.4 (0.7) | 3.5 (0.6)

ADVERSE EVENTS:
Time Frame: Between baseline assessment through our 24-week postpartum follow-up. This varied across study participants, but generally was approximately 12 months.
Description: We used the clinicaltrials.gov definition of an adverse event. All-Cause Mortality and Serious Adverse Events were not monitored/assessed.
Arm/Group | Mothers and Babies Groups Home-Visitor | Mothers and Babies Groups Clinician | Control
All-Cause Mortality (participants affected / at risk) | 0/405 | 0/310 | 0/159
Serious Adverse Events (participants affected / at risk) | 0/405 | 0/310 | 0/159
Other Adverse Events (participants affected / at risk) | 0/405 | 0/310 | 0/159

LIMITATIONS AND CAVEATS:
Our overall sample's baseline depressive symptom score falls in the mild symptom range of the QIDS. There may have been a potential flooring effect in which there was less room to demonstrate improvement in symptom reduction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT02979444/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT02979444/SAP_001.pdf